CLINICAL TRIAL: NCT03630120
Title: Adaptive Tyrosine Kinase Inhibitor Therapy In Patients With Advanced Progressive Thyroid Cancer
Brief Title: Adaptive Tyrosine Kinase Inhibitor (TKI) Therapy In Patients With Thyroid Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCC-19442
Record Dates: First submitted 2018-08-10; First posted 2018-08-14 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Thyroid Cancer; Thyroid Cancer, Medullary; Differentiated Thyroid Cancer; Papillary Thyroid Cancer; Follicular Thyroid Cancer; Poorly Differentiated Thyroid Gland Carcinoma
Keywords: Thyroid disease; Tyrosine kinase inhibitor; TKI; Medullary thyroid cancer; DTC; Advanced thyroid cancer; Progressive thyroid cancer; MTC
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid cancer, medullary; Thyroid Cancer, Papillary; Adenocarcinoma, Follicular; Thyroid Diseases; Carcinoma, Medullary | interventions — lenvatinib; Sorafenib; cabozantinib; vandetanib

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Researchers consenting the patients will become unblinded upon treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Standard of Care: DTC (Active Comparator): Standard of Care (SOC) TKI Therapy for Differentiated Thyroid Cancer (DTC): Lenvatinib + Sorafenib.
  Interventions: Drug: Lenvatinib; Drug: Sorafenib
- Adaptive Care: DTC (Experimental): SOC followed by Adaptive Care TKI Therapy for DTC Participants with >=50% drop: Lenvatinib + Sorafenib.
  Interventions: Drug: Lenvatinib; Drug: Sorafenib
- Standard of Care: MTC (Active Comparator): Standard of Care (SOC) TKI Therapy for Medullary Thyroid Cancer: Cabozantinib + Vandetanib.
  Interventions: Drug: Cabozantinib; Drug: Vandetanib
- Adaptive Care: MTC (Experimental): SOC followed by Adaptive Care TKI Therapy for MTC Participants with >=50% drop: Cabozantinib + Vandetanib.
  Interventions: Drug: Cabozantinib; Drug: Vandetanib

INTERVENTIONS:
Drug: Lenvatinib — Standard of Care: Lenvatinib 24 mg daily. All participants will start receiving standard of care treatment.
  Participants in the Adaptive Therapy regimen will receive TKI therapy in cycles: continuous treatment at the indicated dose until the patients' tumor marker (thyroglobulin in DTC or calcitonin in MTC patients) drops by ≥50% from the level at the time of enrollment ("baseline" level). A new cycle of TKI treatment will begin when/if the tumor marker increases to or above the "baseline" level.
  Other Names: Lenvima®
  Arms: Adaptive Care: DTC; Standard of Care: DTC
Drug: Sorafenib — Standard of Care: Sorafenib 400 mg twice daily. All participants will start receiving standard of care treatment.
  Participants in the Adaptive Therapy regimen will receive TKI therapy in cycles: continuous treatment at the indicated dose until the patients' tumor marker (thyroglobulin in DTC or calcitonin in MTC patients) drops by ≥50% from the level at the time of enrollment ("baseline" level). A new cycle of TKI treatment will begin when/if the tumor marker increases to or above the "baseline" level.
  Other Names: Nexavar®
  Arms: Adaptive Care: DTC; Standard of Care: DTC
Drug: Cabozantinib — Standard of Care: Cabozantinib 140 mg daily. All participants will start receiving standard of care treatment.
  Participants in the Adaptive Therapy regimen will receive TKI therapy in cycles: continuous treatment at the indicated dose until the patients' tumor marker (thyroglobulin in DTC or calcitonin in MTC patients) drops by ≥50% from the level at the time of enrollment ("baseline" level). A new cycle of TKI treatment will begin when/if the tumor marker increases to or above the "baseline" level.
  Other Names: Cabometyx®
  Arms: Adaptive Care: MTC; Standard of Care: MTC
Drug: Vandetanib — Standard of Care: Vandetanib 300 mg daily. All participants will start receiving standard of care treatment.
  Participants in the Adaptive Therapy regimen will receive TKI therapy in cycles: continuous treatment at the indicated dose until the patients' tumor marker (thyroglobulin in DTC or calcitonin in MTC patients) drops by ≥50% from the level at the time of enrollment ("baseline" level). A new cycle of TKI treatment will begin when/if the tumor marker increases to or above the "baseline" level.
  Other Names: Caprelsa®
  Arms: Adaptive Care: MTC; Standard of Care: MTC

SUMMARY:
Participants will have been diagnosed with advanced progressive thyroid cancer and are about to start treatment with a tyrosine kinase inhibitor (TKI).

The purpose of this study is to evaluate the efficacy and tolerability of tyrosine kinase inhibitor therapy (Lenvatinib or Sorafenib for differentiated thyroid cancer [which includes papillary thyroid cancer, follicular thyroid cancer, and poorly differentiated thyroid cancer]; and Cabozantinib or Vandetanib for medullary thyroid cancer) through adaptive (intermittent) versus conventional (continuous) regimen.

DETAILED DESCRIPTION:
Population: Patients with advanced progressive 131I-refractory DTC or MTC will be enrolled to this study. Forty-five patients responding to TKI therapy (defined as 50% drop in tumor marker level within the first two months of treatment) will be randomized to receive TKI therapy either through adaptive (intermittent) or conventional (continuous) regimen.

ELIGIBILITY:
Inclusion Criteria:

* All histologically or cytologically confirmed diagnosis of thyroid cancer, other than anaplastic or stromal-cell derived cancers.
* Participants with differentiated thyroid cancers (DTC) must have negative thyroglobulin antibodies.
* Measurable disease meeting the following criteria and confirmed by central radiographic review:

  * At least 1 lesion of ≥ 1.0 centimeter (cm) in the longest diameter for a non- lymph node or ≥ 1.5 cm in the short-axis diameter for a lymph node which is serially measurable according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 using computerized tomography/magnetic resonance imaging (CT/MRI). If there is only one target lesion and it is a non-lymph node, it should have a longest diameter of ≥ 1.5 cm.
  * Lesions that have had external beam radiotherapy (EBRT) or locoregional therapies such as radiofrequency (RF) ablation must show evidence of progressive disease (substantial size increase of ≥ 20%) within 12 months to be deemed a target lesion.
* Participants must show evidence of disease progression comparing (a) scan in screening and (b) historical scan obtained within 12 months prior to signing informed consent, according to RECIST 1.1 assessed and confirmed by central radiographic review of CT and/or MRI scans.
* Participants with DTC must not be eligible for possible curative surgery and must be radioiodine (RAI)-refractory / resistant as defined by at least one of the following:

  * One or more measurable lesions that do not demonstrate iodine uptake on any radioiodine scan
  * One or more measurable lesions that has progressed by RECIST 1.1 within 12 months of RAI therapy, despite demonstration of radioiodine avidity at the time of that treatment by pre- or post-treatment scanning.
  * Disease progression in a patient that has received a cumulative activity of RAI of ≥ 550 millicuries (mCi) (22 gigabecquerels), with the last RAI dose administered at least 6 months prior to study entry.
  * Otherwise deemed not a candidate for further RAI therapy by a multidisciplinary tumor board within 60 days of enrollment.
* Participants with DTC must be receiving thyroxine suppression therapy and thyroid stimulating hormone (TSH) should not be elevated (TSH should be ≤ 0.1 mU/L).
* "Measurable" tumor marker (non-stimulated thyroglobulin >10 ng/mL or CEA>10 ng/ML in patients with DTC; or serum basal calcitonin >10 pg/mL in patients with MTC)
* Participants may have received prior multi-kinase targeted therapy except the TKI used in this trial. For example, patients getting Lenvatinib on this study may have been previously treated with Sorafenib, Vandetanib, Sunitinib, Pazopanib, etc. Each of the TKI targeted agents will be counted individually, regardless of the duration of its administration.
* Participants with known brain metastases who have completed whole brain radiotherapy, stereotactic radiosurgery or complete surgical resection, will be eligible if they have remained clinically stable, asymptomatic for 30 days.
* All chemotherapy or radiation related toxicities must have resolved to < Grade 2 severity per Common Terminology Criteria for Adverse Events (CTCAE v 5.0), except alopecia infertility, anemia (see separate criteria) and any toxicities deemed irreversible by the treating physician.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 - 2.
* Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤ 150/90 mm Hg at screening and no change in antihypertensive medications within 1 week prior to Cycle 1/Day 1
* Adequate renal function defined as calculated creatinine clearance ≥ 30 mL/min (using Cockcroft/Gault formula)
* Adequate bone marrow function
* Adequate liver function
* Males or females age ≥ 18 years at the time of informed consent
* Females must not be breastfeeding or pregnant at Screening or Baseline.
* Males and females must follow all contraception guidelines as outlined in the protocol guidelines.
* Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol

Exclusion Criteria:

* Participants who have received any anticancer treatment (including Chinese herbal medicine specified for the treatment of tumor) within 21 days or any investigational agent within 30 days prior to the first dose of study drug. This does not apply to the use of TSH-suppressive thyroid hormone therapy.
* Major surgery within 21 days prior to the first dose of study drug.
* Palliative radiation therapy within 14 days prior to the first dose of study drug.
* Participants having > 30 mg/mL urine protein on urine dipstick testing (Participants with urine protein < 1 g/24 hour (h) will be eligible).
* Gastrointestinal malabsorption or any other condition that in the opinion of the investigator might affect the absorption of Lenvatinib, Sorafenib, Cabozantinib, or Vandetanib.
* Significant cardiovascular impairment: history of (a) congestive heart failure greater than New York Heart association (NYHA) Class II, (b) unstable angina, (c) myocardial infarction, (d) stroke, or (e) cardiac arrhythmia associated with impairment within 6 months of the first dose of study drug.
* Bleeding or thrombotic disorders (Treatment with low molecular weight heparin is allowed).
* Radiographic evidence of major blood vessel invasion/infiltration.
* Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 21 days prior to the first dose of study drug.
* Active infection (any infection requiring systemic treatment).
* Active malignancy (except for DTC/MTC or definitively treated basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix or bladder) within the past 24 months.
* Known intolerance to any of the study drugs (or any of the excipients).
* Any medical or other condition which, in the opinion of the investigator, would preclude participation in a clinical trial.
* Females who are pregnant or breastfeeding.
* Participants who are taking prohibited medications outlined in protocol documentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine H. Chung, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Adaptive Care: DTC: SOC followed by Adaptive Care TKI Therapy for DTC Participants with >=50% drop: Lenvatinib + Sorafenib.
  Lenvatinib: Standard of Care: Lenvatinib 24 mg daily. All participants will start receiving standard of care treatment.
  Participants in the Adaptive Therapy regimen will receive TKI therapy in cycles: continuous treatment at the indicated dose until the patients' tumor marker (thyroglobulin in DTC or calcitonin in MTC patients) drops by ≥50% from the level at the time of enrollment ("baseline" level). A new cycle of TKI treatment will begin when/if the tumor marker increases to or above the "baseline" level.
  Sorafenib: Standard of Care: Sorafenib 400 mg twice daily. All participants will start receiving standard of care treatment.
  Participants in the Adaptive Therapy regimen will receive TKI therapy in cycles: continuous treatment at the indicated dose until the patients' tumor marker (thyroglobulin in DTC or calcitonin in MTC patients) drops by ≥50% from the level at the time of enrollment ("baseline" level). A new cycle of TKI treatment will begin when/if the tumor marker increases to or above the "baseline" level.
- Adaptive Care: MTC: SOC followed by Adaptive Care TKI Therapy for MTC Participants with >=50% drop: Cabozantinib + Vandetanib.
  Cabozantinib: Standard of Care: Cabozantinib 140 mg daily. All participants will start receiving standard of care treatment.
  Participants in the Adaptive Therapy regimen will receive TKI therapy in cycles: continuous treatment at the indicated dose until the patients' tumor marker (thyroglobulin in DTC or calcitonin in MTC patients) drops by ≥50% from the level at the time of enrollment ("baseline" level). A new cycle of TKI treatment will begin when/if the tumor marker increases to or above the "baseline" level.
  Vandetanib: Standard of Care: Vandetanib 300 mg daily. All participants will start receiving standard of care treatment.
  Participants in the Adaptive Therapy regimen will receive TKI therapy in cycles: continuous treatment at the indicated dose until the patients' tumor marker (thyroglobulin in DTC or calcitonin in MTC patients) drops by ≥50% from the level at the time of enrollment ("baseline" level). A new cycle of TKI treatment will begin when/if the tumor marker increases to or above the "baseline" level.
Period: Overall Study
Arm/Group | Standard of Care: DTC | Adaptive Care: DTC | Standard of Care: MTC | Adaptive Care: MTC
Started | 2 | 2 | 1 | 1
Completed | 2 | 1 | 0 | 0
Not Completed | 0 | 1 | 1 | 1
Not completed — Disease progression | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care: DTC: Standard of Care (SOC) TKI Therapy for Differentiated Thyroid Cancer (DTC): Lenvatinib + Sorafenib.
  Lenvatinib: Standard of Care: Lenvatinib 24 mg daily. All participants will start receiving standard of care treatment.
  Participants in the Adaptive Therapy regimen will receive TKI therapy in cycles: continuous treatment at the indicated dose until the patients' tumor marker (thyroglobulin in DTC or calcitonin in MTC patients) drops by ≥50% from the level at the time of enrollment ("baseline" level). A new cycle of TKI treatment will begin when/if the tumor marker increases to or above the "baseline" level.
  Sorafenib: Standard of Care: Sorafenib 400 mg twice daily. All participants will start receiving standard of care treatment.
  Participants in the Adaptive Therapy regimen will receive TKI therapy in cycles: continuous treatment at the indicated dose until the patients' tumor marker (thyroglobulin in DTC or calcitonin in MTC patients) drops by ≥50% from the level at the time of enrollment ("baseline" level). A new cycle of TKI treatment will begin when/if the tumor marker increases to or above the "baseline" level.
- Standard of Care: MTC: Standard of Care (SOC) TKI Therapy for Medullary Thyroid Cancer: Cabozantinib + Vandetanib.
  Cabozantinib: Standard of Care: Cabozantinib 140 mg daily. All participants will start receiving standard of care treatment.
  Participants in the Adaptive Therapy regimen will receive TKI therapy in cycles: continuous treatment at the indicated dose until the patients' tumor marker (thyroglobulin in DTC or calcitonin in MTC patients) drops by ≥50% from the level at the time of enrollment ("baseline" level). A new cycle of TKI treatment will begin when/if the tumor marker increases to or above the "baseline" level.
  Vandetanib: Standard of Care: Vandetanib 300 mg daily. All participants will start receiving standard of care treatment.
  Participants in the Adaptive Therapy regimen will receive TKI therapy in cycles: continuous treatment at the indicated dose until the patients' tumor marker (thyroglobulin in DTC or calcitonin in MTC patients) drops by ≥50% from the level at the time of enrollment ("baseline" level). A new cycle of TKI treatment will begin when/if the tumor marker increases to or above the "baseline" level.
- Total: Total of all reporting groups
Arm/Group | Standard of Care: DTC | Adaptive Care: DTC | Standard of Care: MTC | Adaptive Care: MTC | Total
Number analyzed (Participants) | 2 | 2 | 1 | 1 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 1 | 4
  >=65 years | 1 | 1 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1 | 2
  Male | 2 | 2 | 0 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 2 | 1 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 1 | 1 | 6
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 1 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Time to Tyrosine Kinase Inhibitor (TKI) Treatment Discontinuation Due to Progressive Disease
Description: Median time-to-discontinuation (TTD) of treatment per study arm, due to Progressive Disease.
Time Frame: 2 years
Population: Data not collected. Only 3 participants remained on study treatment, and none for full length of trial.
Arm/Group | Standard of Care: DTC | Adaptive Care: DTC | Standard of Care: MTC | Adaptive Care: MTC
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Time to Tyrosine Kinase Inhibitor (TKI) Treatment Discontinuation Due to Intolerability
Description: Median time-to-discontinuation (TTD) of treatment per study arm, due to Intolerability.
Time Frame: 2 years
Population: Data not collected. Only 3 participants remained on study treatment, and none for full length of trial.
Arm/Group | Standard of Care: DTC | Adaptive Care: DTC | Standard of Care: MTC | Adaptive Care: MTC
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Primary Outcome: Time to Tyrosine Kinase Inhibitor (TKI) Treatment Discontinuation Due to Disease Related Death
Description: Median time-to-discontinuation (TTD) of treatment per study arm, due to Disease-related death at 2 years.
Time Frame: 2 years
Population: Data not collected. Only 3 participants remained on study treatment, and none for full length of trial.
Arm/Group | Standard of Care: DTC | Adaptive Care: DTC | Standard of Care: MTC | Adaptive Care: MTC
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Overall Response Rate (ORR)
Description: The response rate will be estimated using binomial theory with Wilson's method for the 95% confidence interval. Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter (LD). Stable Disease (SD): Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum LD since the treatment started.
Time Frame: Up to 48 months
Population: Data not collected. Only 3 participants remained on study treatment, and none for full length of trial.
Arm/Group | Standard of Care: DTC | Adaptive Care: DTC | Standard of Care: MTC | Adaptive Care: MTC
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Progression-free Survival (PFS)
Description: The median progression-free survival rates will be estimated from the Kaplan-Meier curve with the 95% confidence interval obtained from Greenwood's formula. Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Up to 48 months
Population: Data not collected. Only 3 participants remained on study treatment, and none for full length of trial.
Arm/Group | Standard of Care: DTC | Adaptive Care: DTC | Standard of Care: MTC | Adaptive Care: MTC
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Overall Survival (OS)
Description: The median overall survival rates will be estimated from the Kaplan-Meier curve with the 95% confidence interval obtained from Greenwood's formula.
Time Frame: Up to 48 months
Population: Data not collected. Only 3 participants remained on study treatment, and none for full length of trial.
Arm/Group | Standard of Care: DTC | Adaptive Care: DTC | Standard of Care: MTC | Adaptive Care: MTC
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year, 4 months
Arm/Group | Standard of Care: DTC | Adaptive Care: DTC | Standard of Care: MTC | Adaptive Care: MTC
All-Cause Mortality (participants affected / at risk) | 0/2 | 1/2 | 1/1 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 0/2 | 0/1 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care: DTC (N=2) | Adaptive Care: DTC (N=2) | Standard of Care: MTC (N=1) | Adaptive Care: MTC (N=1)
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT03630120/Prot_SAP_000.pdf